CLINICAL TRIAL: NCT00766896
Title: Platelet Hyperreactivity to Aspirin and Stroke: A Prospective Study With Clinical Outcomes
Brief Title: Platelet Hyperreactivity to Aspirin and Stroke
Acronym: PLARAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Accumetrics, Inc. (Industry); Helena Laboratories Point of Care (Unknown); Chrono-Log Corporation (Unknown)
Responsible Party: Principal Investigator, Herlon Saraiva Martins, Herlon Saraiva Martins, M.D., Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 0292/07
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Stroke; Cerebral Infarction; Cardiovascular Diseases; Vascular Diseases; Atherosclerosis; Ischemia; Thrombosis; Acute Coronary Syndrome
Keywords: Stroke; Cerebral Infarction; Acute Coronary Syndrome; Cardiovascular Diseases; Vascular Diseases; Platelet Activation; Platelets; Platelet Function Tests; Aspirin; Atherosclerosis; Ischemia; Thrombosis
MeSH Terms: conditions — Stroke; Cerebral Infarction; Cardiovascular Diseases; Vascular Diseases; Atherosclerosis; Ischemia; Thrombosis; Acute Coronary Syndrome | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin Sensitive (Active Comparator): * For PFA-100 using a cartridge with C-EPI (collagen-epinephrine): occlusion time >= 150 seconds
  * Chrono-Log Model 700 Whole-Blood: < 1Ω with 0.75 mM of arachidonic acid
  * Chrono-Log Model 700 Whole-Blood: with collagen at 1 mg/L and 5 mg/L, according to the formula 1 - (Rate of aggregation with 1 mg / Rate of aggregation with 5 mg) > 0.50
  * Chrono-Log Model 700 Whole-Blood: with collagen at 1 mg/L < 10Ω
  * Plateletworks: aggregation <60% with arachidonic acid will be considered sensitive
  * VerifyNow Aspirin Assay (Accumetrics): < 550 aspirin reaction units (ARUs)
  * Impact-R (Diamed) < 3.2% platelet aggregates on the surface of the plate after incubation with arachidonic acid
  Interventions: Drug: Aspirin (platelet sensitive versus platelet hyperreactivity)
- Platelet with hyperreactivity to aspirin (Active Comparator): * For PFA-100 using a cartridge with C-EPI (collagen-epinephrine): occlusion time < 150 s
  * Chrono-Log Whole-Blood: above or = 1Ω with 0.75 mM of AA
  * Chrono-Log Whole-Blood: with collagen at 1 mg/L and 5 mg/L, according to the formula 1 - (Rate of aggregation with 1 mg / Rate of aggregation with 5 mg) below 0.50
  * Chrono-Log Whole-Blood: with collagen 1 mg/L above or = 10Ω
  * Plateletworks: aggregation of more than 60% with arachidonic acid will be considered resistant
  * VerifyNow Aspirin Assay (Accumetrics): ≥ 550 aspirin reaction units (ARUs)
  * Impact-R (Diamed) > 3.2% platelet aggregates on the surface of the plate after incubation with arachidonic acid
  Interventions: Drug: Aspirin (platelet sensitive versus platelet hyperreactivity)

INTERVENTIONS:
Drug: Aspirin (platelet sensitive versus platelet hyperreactivity) — The dose of aspirin to be prescribed in this study will be 300 mg orally or by nasogastric tube once a day (assisted therapy), with first dose tomography soon after admission if the patient has no indication of thrombolytic therapy. After the acute phase, patients will receive aspirin at a dose of 200 mg/day. Aspirin will be administered in a "simple" preparation (no buffer, no extended release).
  Other Names: Aspirin resistance

SUMMARY:
STUDY QUESTIONS

* What is the real prevalence of platelet "resistance" to aspirin during the acute phase of stroke and after 3 months, and 1 year, as measured using different platelet function tests?
* Do all methods measure similar levels of resistance, or are some methods more sensitive than others?
* Does this resistance result in a worse clinical prognosis? Is this result independent of other variables?

OBJECTIVES

1. Hospital Phase (Acute Stroke)

   * Determination, using various methods, of the prevalence of platelet hyperreactivity in patients treated with aspirin to treat ischemic stroke (acute phase)
   * Comparison of different assessment methods and identification of the most accurate of these
   * Identification of variables that correlate with platelet hyperreactivity
2. Follow-up Phase

   * Correlation between platelet hyperreactivity and important clinical outcomes at 12, 24, and 36 months
   * Correlation between platelet hyperreactivity and death or dependency at hospital discharge, at 3, 12, 24, and 36 months (Modified Rankin Scale)
   * Correlation between platelet hyperreactivity and recurrent stroke of any type
   * Correlation between different methods for evaluating platelet functions and identification of the most accurate method
   * Analysis of hyperreactivity over time

THE STUDY

* The study will include 200 consecutive patients seen in the emergency department of a large, urban hospital (1500 inpatient beds) and diagnosed with stroke in the acute phase; these patients will be treated with aspirin for an undetermined period
* The investigators will not include patients who require full anticoagulation treatment, regardless of the cause
* Importantly, the analysis of primary and secondary outcomes will be carried out after blinding the examiner to the results of the platelet aggregation tests

PLATELET TESTS

* Whole Blood Aggregometer, ChronoLog
* VerifyNow, Accumetrics
* PFA-100, Siemens
* Plateletworks, Helena
* Impact-R, Diamed
* Serum thromboxane B2

DETAILED DESCRIPTION:
THE CONTEXT

Aspirin is the anti-thrombotic therapy of choice for patients in the acute or chronic phase of vascular, cardiac, and neurological diseases, unless there is a specific indication for sodium warfarin (for instance, cardiac thrombus, chronic atrial fibrillation, cardio-embolic ischemic stroke). Recent studies, including some meta-analyses, suggest that 5-60% of patients with cardiovascular disease who use aspirin show some platelet resistance to the drug. However, the available studies include several methodological errors that make interpretation and practical application difficult. Thus, the incidence and outcome of platelet resistance remain poorly understood, especially in patients with ischemic stroke. Moreover, few studies have included patients in ambulatory follow-up

THERAPY WITH ASPIRIN

The dose of aspirin to be prescribed in this study will be 300 mg orally or by nasogastric tube once a day (assisted therapy), with first dose tomography soon after admission if the patient has no indication of thrombolytic therapy. After the acute phase, patients will receive aspirin at a dose of 200 mg/day. Aspirin will be administered in a "simple" preparation (no buffer, no extended release)

ANALYSIS OF OUTCOME DURING THE HOSPITAL PHASE

The outcomes will be assessed daily during hospitalization until the patient is discharged. The physician, the patient, and the researchers will not have access to the results of tests for platelet function. The number of days of hospitalization will be reviewed, including the number of days of hospitalization in the intensive care unit. Deaths will be analyzed, and the cause of death will be described in detail in each case. Electrocardiograms will be examined by an experienced cardiologist. Echocardiograms will be examined by an experienced cardiologist specializing in this method. Tomography will be examined by an experienced neuroradiologist, and resonance/resonance angiography will be evaluated by another experienced neuroradiologist; both will be blinded to the platelet results. Outcomes will be judged by a committee containing a neurologist, a hematologist, a neuroradiologist, a cardiologist, and an epidemiologist, all of whom will be blinded to the results of platelet function

MONITORING AND MANAGEMENT AFTER HOSPITAL DISCHARGE

Outcomes will be analyzed through interviews 3, 12, 24, and 36 months after the initial neurological event, as well as with monthly telephone interviews. Potential adverse outcomes (death, hospitalization, diagnostic tests conducted, request for treatment of any condition, or new onset of symptoms) will be assessed in detail by the committee of investigators of this study. During this evaluation, the doctor, the patient, and the researchers will not have access to the results of the tests for platelet function. The outcomes will be judged by a committee comprising a neurologist, a hematologist, a neuroradiologist, a cardiologist, and an epidemiologist, all of whom will be blinded to platelet test results Adherence (daily use) will be investigated in an active manner at all return visits and through monthly telephone contact. This study will include interviews with patients and separate interviews with families, in addition to reviews of the package of aspirin. In addition, adherence will be assessed by measuring serum thromboxane B2.

* Monthly telephone contact with the patient and his or her family will be used to determine whether the patient has remained stable or has had any adverse outcome (died, needed to seek medical care, or presented new symptoms). In the presence of any such outcomes, we will investigate the details (death certificate, report of hospital stay, and analysis of diagnostic tests performed). In addition, we will investigate the records and medical reports associated with any inquiries or admissions.
* The evaluation at three and twelve months will consist of a variety of tests of platelet function; in addition, a standardized questionnaire will be administered. Patients who do not attend the consultation will be contacted within 30 days. If the patient still cannot attend the consultation (e.g., because of difficulty in walking), the researcher will go to the patient's home.

SEVERE BLEEDING

* Any fatal bleeding event (all causes will be described)
* Life-threatening bleeding: a drop in hemoglobin of at least 50 g/L, hypotension requiring inotropes (hemorrhagic shock); symptomatic intracranial hemorrhage; or transfusion of at least 4 units of red blood cells
* Major bleeding, defined as significantly disabling (with persistent sequelae); intraocular bleeding leading to significant loss of vision; or transfusion of 1-3 units of red blood cells

DEFINITION OF HYPERREACTIVITY TO ASPIRIN

* For PFA-100 using a cartridge with C-EPI (collagen-epinephrine): occlusion time < 150 seconds
* Chrono-Log Model 700 Whole-Blood: above 0 Ω with 0.75 mM of arachidonic acid
* Chrono-Log Model 700 Whole-Blood: with collagen at 1 mg/L and 5 mg/L, according to the formula 1 - (Rate of aggregation with 1 mg / Rate of aggregation with 5 mg). Hyperreactivity will be defined for values below 0.50
* - Chrono-Log Model 700 Whole-Blood: with collagen at 1 mg/L above 10 Ω
* Plateletworks: aggregation of more than 60% with arachidonic acid will be considered resistant
* VerifyNow Aspirin Assay (Accumetrics): ≥ 550 aspirin reaction units (ARUs)
* Impact-R (Diamed) > 3.2% platelet aggregates on the surface of the plate after incubation with arachidonic acid

COLLECTION OF BLOOD

Blood samples will be collected on arrival at the ED (before the first dose of aspirin), on the fifth day of hospitalization, after three months, and again after 12 months. Samples will be collected between 9 and 12 AM after fasting overnight, except for the sample taken on arrival at the ED. The blood will be collected from the antecubital vein, or another vein if necessary, into bottles of citrate (3.2%; Vacuette, Greiner Bio-One) or directly into the Plateletworks bottle kit. Samples will total approximately 20 ml. The tourniquet will not be applied for more than 30 seconds and movement will not be allowed before or during collection. In order to prevent platelet activation induced by collection, even with the above precautions, the first 5 ml sample will be discarded. The bottles will be filled to the top and gently inverted five times to obtain the correct mixture of blood with anticoagulant. In the Plateletworks test, assays will conducted within 10 minutes of collection; the remaining assays will be conducted within 30 minutes

AGGREGOMETRY BY MEASURING THE IMPEDANCE OF WHOLE BLOOD USING CHRONOLOG MODEL 700 AND SOFTWARE (AGGRO/LINK-8, PA, USA)

After collecting citrated whole blood, the sample will be processed in under 30 minutes. Whole blood will be diluted 1:1 with sterile saline (0.9%) and stimulated with one of several reagents (Chrono-Log, 0.5 mM arachidonic acid, 1 g/L collagen, or 5 g/L collagen). The maximum impedance will be measured using two electrodes immersed in the sample for 6 minutes and expressed as Ω.

PFA-100 (PLATELET FUNCTION ANALYZE-100, SIEMENS, USA)

Blood specimens for PFA-100® assays will be tested according to the manufacturer's instructions. For all samples, the PFA-100® self-test procedure will be run before analysis. Testing will be performed using citrated whole blood with collagen-epinephrine cartridges. Whole blood will be aspirated under conditions of high shear stress through a 150-µm aperture covered with a membrane impregnated with collagen and epinephrine. The time taken to occlude the aperture by a platelet plug will be recorded as the closure time (measured in seconds).

DETERMINATION OF SERUM THROMBOXANE B2 - ELISA

After collection, blood will be immediately centrifuged (+4 °C), and the plasma immediately frozen in liquid nitrogen (-190 °C) and then transferred to a -80 °C freezer. Serum thromboxane B2 will be measured by ELISA in duplicate according to the manufacturer's instructions, and expressed as ng/ml.

PLATELETWORKS (HELENA CORPORATION, USA)

Briefly, after collection of blood in kits containing arachidonic acid, collagen, ADP and EDTA, platelet counts will be made by impedance measurement (Horiba ABX, Montpellier, France), in accordance with the standard protocol of Helena Laboratories (Helena Point of Care ®, Texas, USA). The percentage of platelet aggregation will be calculated using the following formula: % of aggregation = [platelets in EDTA - platelets with agonist]/ platelets in EDTA x 100

VERIFYNOW ASPIRIN, ACCUMETRICS, USA

The VerifyNow Aspirin point-of-care system (Accumetrics, San Diego, CA, USA) is based on turbidimetric optical detection of platelet aggregation in whole blood. Whole blood will be transferred into standard cartridges containing a lyophilized preparation of human fibrinogen-coated beads and arachidonic acid. As aggregation occurs, the system will convert luminosity transmittance results into aspirin reaction units (ARUs).

IMPACT-R, DIAMED, USA

Citrated blood (130 μL) will be placed in the test kit (wells) according to the manufacturer's protocol, and subjected to shear flow using a rotating cone for 2 minutes (1800 s-1). The wells will then be washed and stained with May Grünwald. The adhesion of platelets to the surface will be evaluated using an image analysis system connected to the Impact-R, and the results will be expressed as the percentage of stained area.

STATISTICAL ANALYSIS

For all calculations, will be used the software IBM SPSS 21.0 for Windows (SPSS Inc, Chicago, IL, USA). The database will be created by SPSS Data Entry Builder 4.0 using the double entry input system.

TIMETABLE FOR IMPLEMENTATION OF THE PROJECT

Phase No. of Months Calendar Dates Trial Activities and Estimates

1. 13 03/2007 - 04/2008 Protocol Development
2. 2 05/2008 - 06/2008 Procedure Finalization
3. 5 07/2008 - 12/2008 Protocol Revision
4. 6 01/2009- 06/2009 Training
5. 12 07/2009 - 06/2010 Main trial recruitment in emergency room
6. 36 08/2009 - 06/2013 Follow-up
7. 3 07/2013 - 10/2013 Analysis and reporting.

CONFLICT OF INTEREST

There is no external influence or sponsor for the survey, collection, or analysis of data. Similarly, the statistical analysis, preparation and publication of manuscripts will be conducted entirely by the researchers themselves, working together with epidemiologists and statisticians of the Faculty of Medicine, USP. Companies and institutions that provided the kits and equipment for the platelet tests will be described in presentations at conferences and in publications

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with the diagnosis of ischemic stroke in the acute phase who will be treated with aspirin for an indefinite period

Exclusion Criteria:

* The need for full anticoagulation therapy for pulmonary embolism, deep vein thrombosis, chronic atrial fibrillation, thrombus in the left atrium or left ventricle, or for any other reason deemed relevant by the patient's physician
* Thrombolytic treatment for stroke
* History of allergy to aspirin (hives, swelling of glottis or anaphylaxis)
* Risk of excessive bleeding due to active peptic ulcers, liver failure, history of bleeding or bleeding diathesis
* Scheduled major or vascular surgery
* Metastatic cancer or survival estimated at less than a year
* Creatinine clearance below 30 mL/min
* Platelet count <100,000/mm3
* Hematocrit <30%
* Lipaemic blood
* Difficult follow-up: patients with serious social problems, alcoholics, and residents of other states in the country
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Correlation between platelet hyperreactivity and the sum of clinical outcomes (sum of death, TIA, stroke and acute coronary syndromes) in 3, 12, 24, and 36 months | Three, 12, 24, and 36 months

SECONDARY OUTCOMES:
Primary outcomes for subgroups [(a) recent use of aspirin, (b) TOAST (c) SSS-TOAST] | Three, 12, 24, 36 months
Compare TOAST with SSS-TOAST | During the initial hospitalization
Severe bleeding | Three, 12, 24, 36 months
Prevalence, correlation and accuracy of various tests of platelet function | Three, 12, 24, 36 months
Correlation between platelet hyperreactivity and the clinical outcomes individually (TIA and stroke; acute coronary syndromes; death) | Three, 12, 24, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Herlon S Martins, MD, Study Chair — University of Sao Paulo, Hospital das Clinicas, Department of Emergency Medicine; Irineu T Velasco, PHD, Study Chair — University of Sao Paulo, Hospital das Clínicas, Department of Emergency Medicine; Élbio A D'Amico, PHD, Study Director — University of Sao Paulo, Hospital das Clínicas, Department of Hematology; Tânia RF Rocha, PHD, Principal Investigator — University of Sao Paulo, Hospital das Clínicas, Department of Hematology; Moacyr RC Nobre, PHD, Study Director — University of Sao Paulo, Unidade de Epidemiologia Clínica; Luíz R Comerlatti, MD, Principal Investigator — University of Sao Paulo, Hospital das Clínicas, Department of Neurology; Cláudia C Leite, PHD, Study Director — University of Sao Paulo, Hospital das Clínicas, Department of Radiology; José L Andrade, MD, Study Director — University of Sao Paulo, Hospital das Clínicas, Department of Radiology
Locations (1):
- University of Sao Paulo, School of Medicine, São Paulo, São Paulo, Brazil